CLINICAL TRIAL: NCT00943748
Title: Efficacy and Safety of the Iron Chelator Deferiprone on Iron Overload in the Brain in Parkinson's Disease
Brief Title: Efficacy and Safety of the Iron Chelator Deferiprone in Parkinson's Disease
Acronym: FAIR-PARK-I
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2008-006842-25; 2008_19/0838 (Other: sponsor); A90113-62 (Other: AFSSAPS)
Record Dates: First submitted 2009-07-20; First posted 2009-07-22 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2009-07

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease | interventions — Deferiprone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- deferiprone (Active Comparator): deferiprone 30 mg/kg/day
  Interventions: Drug: deferiprone
- placebo (Placebo Comparator): placebo : 30 mg/kg/day, in 2 liquid doses
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: deferiprone — A standard dose-escalation phase will be initiated, with a 3 ml of the deferiprone oral solution twice a day (breakfast and dinner) increase every 3 days up to a total of a fixed dose of 9 ml of deferiprone oral solution twice a day corresponding to 30 mg/kg/day in 2 doses
  Other Names: FERRIPROX
  Arms: deferiprone
Drug: placebo — A standard dose-escalation phase will first be initiated, with a 3 ml of the placebo oral solution twice a day (breakfast and dinner) increase every 3 days up to a total of a fixed dose of 9 ml of placebo oral solution twice a day corresponding to 30 mg/kg/day in 2 doses
  Arms: placebo

SUMMARY:
Few available drugs can slow the progression of neurodegenerative pathologies such as Parkinson's disease (PD). One of the recent hypotheses concerning the reduction of oxidative stress and neuron death features a harmful effect of iron, which may reach abnormally high levels in the substantia nigra (SN) pars compacta (iron overload has been seen in the substantia nigra in parkinsonian patients and in the 1-methyl-4-phenyl-1,2,3,6-tetrahydropyridine (MPTP) mouse model of PD). Iron overload is harmful because it reacts with hydrogen peroxide (H2O2) produced during the oxidative deamination of dopamine, generating hydroxyl radicals which then damage proteins, DNA and phospholipid membranes and may be responsible for neuron death. The use of an iron chelator (clioquinol) produces a reduction in neuron death in the MPTP mouse model. In humans, a special, partially refocused interleaved multiple echo (PRIME) MR sequence has been used to study the relaxation time (T2*) and quantify iron overload in the SN of PD patients and the nucleus dentatus of patients with Friedreich's ataxia. T2* sequences have revealed a decrease in iron overload following treatment with the chelator deferiprone, in parallel with a clinical improvement in these patients. Furthermore, the very recent open label use of deferiprone in rare serious, systemic, neurological iron overload diseases (Neurodegeneration with Brain Iron Accumulation (NBIA)) has revealed a clinical improvement after 6 months, with 2 case reports from our group and another from an Italian group (Forni et al., 2008). The safety of the low dosages of deferiprone (20 to 30 mg/kg/day) used in neurology appears to be much greater than for the high dosages (75 to 100 mg/kg/day in 3 doses) used in hematology to decrease post-transfusion iron overloads in thalassemia major.

Hence, the investigators wish to evaluate the effect of treatment with an oral iron chelator which is capable of crossing the blood-brain barrier (deferiprone) on iron overload in the SN(as assessed by the T2* sequence) with respect to the progression of clinical sign in PD. It is expected a 6-month course of deferiprone able to produce a moderate reduction in iron overload of the SN, associated with a drop in the motor handicap score. Depending on the risk/benefit balance determined in this initial pilot study, a larger, multicenter neuroprotection study could be envisaged.

DETAILED DESCRIPTION:
Primary objective: decrease the iron overload (as measured by the T2* MRI sequence) in the substantia nigra in patients with Parkinson's disease (PD) after 6 months of deferiprone treatment, relative to the placebo group.

Secondary objectives:

1. Other radiological criteria: Modification of T2* in MRI of the caudal nucleus head, putamen and pallidum.
2. Evaluate the "disease modifier" effect on the clinical symptoms:

   * Parkinsonian syndrome: UPDRS III
   * the Clinical Global Impression scored by the examiner and the patient.
3. Evaluate the safety on cognitive and behavioral functions

   * MDS-UPDRS I
   * overall cognitive function (Mattis, MMSE), memory, executive function, attention (simple and choice reaction times)
   * drowsiness and sleep (Epworth scale, Parkinson Disease Sleep Scale), depression (MADRS).
4. Safety: complete blood count (CBC) with weekly leukocyte counts, standard blood biochemistry profile, blood iron profile, ECG, blood pressure, bodyweight, adverse event reporting.
5. Specific biochemistry screen: heavy metal profile, oxidative stress and dopamine metabolism.

Study center: Service de Neurologie et Pathologie du Mouvement (Head: Prof. Destée, Clinique Neurologique and Service de Neuroradiologie (Head: Prof. Pruvo), Salengro Hospital, Lille University Medical Center, Lille, France.

Study characteristics: a randomized, double-blind, placebo-controlled, parallel-group, single-center trial with a delayed onset paradigm (Early-start group with 12 months of deferiprone versus delayed -start group with 6 months of placebo then 6 months of deferiprone) to study the effect of deferiprone on the relaxation time of the substantia nigra during a T2* MRI sequence (R2*=1/T2* reflecting iron overload) with respect to motor disorders in Parkinson's disease.

Active compound: the iron chelator 1,2-dimethyl-3-hydroxy-4-pyridinone (deferiprone, FERRIPROX®), which decreases abnormally high iron and ferritin levels. Its low molecular weight and liposolubility enable it to cross the blood-brain barrier.

Posology: the recommended dosage in neurology is a total of 30 mg/kg/day, in 2 doses.

Study population: 40 adult parkinsonian volunteers, with early-stage PD under their first optimised dopaminergic therapeutic strategy (i.e. either dopamine agonist and/or slight dose of L-dopa) and free of motor fluctuations or dementia.

Planned inclusion period: 12 months. Study duration for individual patients: 13 months (2 weeks between screening and randomization, 6 months of double-blind treatment, then 6 months of open label treatment and then a 2-week wash-out period).

Study procedures and timeline:

* A screening visit (Sc).
* Two comprehensive examinations (a neurological and neuropsychological check-up) at the randomization visit (V0, at D7-15 ± 1 week after Sc), visit after 6 months (V6, at least 6 months after V0), visit after 12 months (V12, at least 12 months after V0)
* Weekly monitoring of the CBC with the leukocyte count, results faxed by the patient's local clinical lab or Lille University Medical Center's central lab.
* Monitoring of blood iron and zinc status and overall tolerance during a brief consultation: V1, V3, V5, V7, V9, V11
* MRI in an external facility at V0, V6, V12.
* Telephone follow-up: V2, V4, V8, V10
* Patients will be invited to participate in an ancillary study involving analysis of the cerebrospinal fluid (CSF) at the randomization visit and the V6, in order to perform a full set of CSF biochemistry assays and with a view to determining biological benefits at the central nervous system level and identifying biological markers.

ELIGIBILITY:
Inclusion Criteria:

* Patients with typical Parkinson's disease according to the Gibb criteria and the Parkinson's Disease Society criteria (Daniel and Lees, 1993).
* Ideally less than 2 to 3 years since disease onset and never more than 4 years.
* Patients on dopaminergic drugs and/or L-Dopa.
* Non-fluctuating disease because otherwise the degenerative process would be well advanced, the clinical score would vary from one day to another and the imaging evaluation would be complicated by dyskinesia.

Exclusion Criteria:

* Subjects over the age of 80
* Demented subjects: MMSE score ≤ 24, Mattis score of < 130 and DSM IV criteria
* Subjects with radiological anomalies on MRI, whether incidental or suggestive of vascular involvement or significant cortical or subcortical atrophy
* Subjects for whom MRI is contra-indicated (metal objects in the body, severe claustrophobia, pacemaker, etc.)
* Subjects undergoing brain stimulation
* Very severe rest tremor, which could induce MRI artifacts
* Subjects that have not stabilized in terms of the therapeutic regimen and who are likely to require changes in their dopamine therapy in the coming 6 months
* Hoehn and Yahr stage ≥ 3 in the "Off" state, indicating the need for walking assistance in the absence of treatment.
* Hypersensitivity to iron chelator drugs
* Patients at risk of or having experienced agranulocytosis
* Patients on a drug that can potentially induce agranulocytosis (clozapine, Closaril®/Leponex®)
* Patients with anemia (regardless of the latter's etiology) or a history of other hematological diseases - even an iron deficiency
* Ferritin blood level < 100 ng/ml (100 µg/l)
* A history of hemochromatosis or known iron metabolism disorders.
* Pregnant or breastfeeding women or women not taking effective contraception
* Kidney or liver failure
* Blood coagulation disorders, antiplatelet drugs or anticoagulants
* Concomitant treatment with aluminum-based antacids (interaction)
* Concomitant treatment with vitamin C (interaction)
* Presence of other serious diseases
* Inability to provide informed consent

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-10; Primary Completion 2011-08 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Decrease the iron overload (as measured by the T2* MRI sequence) in the substantia nigra in patients with Parkinson's disease (PD) after 6 months of deferiprone treatment, relative to the placebo group. | 6 months and 12 months

SECONDARY OUTCOMES:
Other radiological criteria: Modification of T2* in MRI of the caudal nucleus head, putamen and pallidum | 6 and 12 months
Parkinsonian syndrome: UPDRS III | 6 and 12 months
Cognitive and behavioral functions: function, attention (simple and choice reaction times), drowsiness and sleep (Epworth scale, Parkinson Disease Sleep Scale), depression (MADRS). | 6 months and 12 months
  MDS-UPDRS I, overall cognitive function (Mattis, MMSE), memory, executive
The Clinical Global Impression scored by the examiner and the patient | 6 months and 12 months
Specific biochemistry screen: heavy metal profile, oxidative stress and dopamine metabolism | 6 and 12 months
Complete blood count (CBC) with weekly leukocyte counts, standard blood biochemistry profile, blood iron profile, ECG, blood pressure, bodyweight, adverse event reporting. | 6 and 12 months
Ancillary study involving analysis of the cerebrospinal fluid (CSF). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: David Devos, MD, PhD, Principal Investigator — Service de Neurologie, Clinique Neurologique, EA 2683, IFR 114, IMPRT
Locations (1):
- Service de Neurologie, Clinique Neurologique, EA 2683, IFR 114, Lille, France

REFERENCES:
- [Derived] Grolez G, Moreau C, Sablonniere B, Garcon G, Devedjian JC, Meguig S, Gele P, Delmaire C, Bordet R, Defebvre L, Cabantchik IZ, Devos D. Ceruloplasmin activity and iron chelation treatment of patients with Parkinson's disease. BMC Neurol. 2015 May 6;15:74. doi: 10.1186/s12883-015-0331-3. PMID 25943368
- [Derived] Devos D, Moreau C, Devedjian JC, Kluza J, Petrault M, Laloux C, Jonneaux A, Ryckewaert G, Garcon G, Rouaix N, Duhamel A, Jissendi P, Dujardin K, Auger F, Ravasi L, Hopes L, Grolez G, Firdaus W, Sablonniere B, Strubi-Vuillaume I, Zahr N, Destee A, Corvol JC, Poltl D, Leist M, Rose C, Defebvre L, Marchetti P, Cabantchik ZI, Bordet R. Targeting chelatable iron as a therapeutic modality in Parkinson's disease. Antioxid Redox Signal. 2014 Jul 10;21(2):195-210. doi: 10.1089/ars.2013.5593. Epub 2014 Feb 6. PMID 24251381